CLINICAL TRIAL: NCT01392846
Title: Evaluation of Effectiveness and Safety of Resolute Integrity DES in Routine Clinical Practice; A Multicenter Prospective Observational Cohort Study (IRIS-Integrity)
Brief Title: The IRIS-Resolute Integrity (IRIS-Integrity)
Status: Completed | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other); Medtronic (Industry)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD,PhD, Chairman,Heart Institute, Asan Medical Center,University of Ulsan,College of Medicine, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Other Study IDs: CVRF2011-07
Record Dates: First submitted 2011-07-11; First posted 2011-07-13 (Estimated); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease requiring drug eluting stents
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Resolute Integrity: Patients receiving Resolute-Integrity stent

SUMMARY:
This is a prospective, observational, cohort study to evaluate the relative efficacy and safety of Resolute Integrity stent compared to other (drug eluting stents) DES.

DETAILED DESCRIPTION:
Consecutive Percutaneous Coronary Intervention patients receiving Resolute Integrity stent will be compared with other concurrent Drug Eluting Stents.

ELIGIBILITY:
Inclusion Criteria:

* Patients with significant coronary artery disease and receiving Resolute Integrity stent.
* The patient or guardian agrees to the study protocol and the schedule of clinical follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethics Committee of the respective clinical site.

Exclusion Criteria:

* Patients with a mixture of other DESs
* Terminal illness with life expectancy <1 year
* Patients presented with cardiogenic shock

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with coronary artery disease requiring drug eluting stents
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2011-07; Primary Completion 2016-01-20 (Actual); Study Completion 2020-03-02 (Actual)

PRIMARY OUTCOMES:
composite of death, nonfatal myocardial infarction (MI), or target- Vessel Revascularization (TVR) | 12 months post procedure

SECONDARY OUTCOMES:
Death (all cause and cardiac) | one month
Death (all cause and cardiac) | 6 months
Death (all cause and cardiac) | 12 months and yearly up to 5 years
Myocardial Infarction | one month
Myocardial Infarction | 6 months
Myocardial Infarction | 12 months and yearly upto 5 years
Composite of death or MI | one month
Composite of death or MI | 6 months
Composite of death or MI | 12 months and yearly upto 5 years
Composite of cardiac death or MI | one month
Composite of cardiac death or MI | 6 months
Composite of cardiac death or MI | 12 months and yearly up to 5 years
Target Vessel Revascularization | one month
Target Vessel Revascularization | 6 months
Target Vessel Revascularization | 12 months and yearly up to 5 years
Target-lesion revascularization | one month
Target-lesion revascularization | 6 months
Target-lesion revascularization | 12 months and yearly up to 5 years
Stent thrombosis | one month
Stent thrombosis | 6 months
Stent thrombosis | 12 months and yearly up to 5 years
Stroke | 12 months and yearly up to 5 years
Procedural success | at day 1
  It is defined as achievement of a final diameter stenosis of <30% by visual estimation, without the occurrence of death, Q-wave MI, or urgent revascularization during the index hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Asan Medical Center
Locations (23):
- South Korea (23):
  - Inje University Ilsan Paik Hospital, Ilsan, Gyeonggi-do
  - Hallym University Sacred Heart Hospital, Anyang
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - The Catholic University of Korea, Bucheon ST.Mary's Hospital, Bucheon-si
  - Soon Chun Hyang University Hospital Cheonan, Cheonan
  - Daegu Catholic University Medical Center, Daegu
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - The Catholic University of Korea, Daejeon ST.Mary's Hospital, Daejeon
  - Gang Neung Asan Hospital, Gangneung
  - Chonnam National University Hospital, Gwangju
  - National Health Insurance Corporation Ilsan Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - Presbyterian Medical Center, Jeonju
  - Kwangju Christian Hospital, Kwangju
  - Pusan National University Yangsan Hospital, Pusan
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Kangdong Sacred Heart Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - St.carollo Hospital, Suncheon
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan